CLINICAL TRIAL: NCT06720649
Title: Benefits of Ballistic Tests in the Decision to Return to Sport After the Ruptured Anterior Cruciate Ligament Surgery
Brief Title: Benefits of Ballistic Tests After the Anterior Cruciate Ligament Surgery
Acronym: BALLCA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Almaviva Sante (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-03; ID-RCB number: 2024-A01538-39 (Other: ANSM)
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patient underwent ACL reconstruction (Experimental)
  Interventions: Other: isokinetic test; Other: Ballistic test; Other: K-STARTS test; Other: Questionnaires

INTERVENTIONS:
Other: isokinetic test — Bilateral strength will be measured using a Contrex ® dynamometer equipped with an exercise table. Each subject will perform isokinetic tests of the right and left knee extensors and flexors. Subjects will be stabilized by straps during testing and the joint rotation axis will be aligned with the input shaft of the dynamometer.
Other: Ballistic test — ballistic squat jumps performed in the supine position on a frictionless sled at a resistance between 0% of body weight (BW)
Other: K-STARTS test — The K-STARTS (Knee Health Athletic Return To Sport) test brings together a set of 7 tests validated in the scientific literature to assess the control and neuromuscular capacities of the lower limb when performing dynamic movements as well as apprehension when resuming activity.
  Test in 30 minutes with physical exercises and questionnaire.
Other: Questionnaires — KOOS (Knee Injury and Osteoarthritis Outcome Score) Questionnaire

SUMMARY:
During physical activities, the time available to produce a force is infinitely shorter than the time required to reach maximal muscle capacity.

Previous studies have observed that the time elapsed between ground contact and ACL rupture is on average 50-60 ms, suggesting that this is the time window available for any attempt at dynamic stabilization of the joint through muscle contraction.

Sports movements include ballistic movements, defined as very fast movements whose objective is to accelerate a moving mass as much as possible so that it reaches a high speed in a very short time. This is the case for vertical jumps, running and most movements performed in physical and sporting activities.

Thus; (1) isokinetic tests do not allow a rigorous analysis of the components related to the speed of the movement; (2) functional tests such as jumping, which only give a distance between one leg and the other, do not allow the calculation of precise and reproducible variables concerning the force and speed of the movement, in particular during the first milliseconds of the movement, and do not provide information on compensation phenomena. It is therefore interesting to use the ballistic tests developed to monitor the movements of athletes as a new possible indicator of the return to sport.

The main objective of this study is to evaluate the performance of ballistic tests in predicting failure to return to physical activity 24 months after ACL surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years),
* Patient who has undergone ACL reconstruction of the hamstrings with or without associated extra-articular plastic surgery:

  * Isolated ACL sprain without injury to the collateral ligaments or the PCL,
  * ACL reconstruction without associated meniscal injury or with repaired or menisctomized meniscal injury,
* Having to perform a K-STARTS test and an isokinetic test,
* Having the Tegner score before the rupture.

Exclusion Criteria:

* Patient with high cardio-respiratory risk,
* Osteoarticular and neuromuscular traumatic sequelae of the lower limbs,
* Degenerative neuromuscular diseases,
* Connective Tissue and Collagen Disease (e.g. Marfan),
* Follow-up of a medical treatment that may influence the neuro-muscular system (e.g., antidepressants, etc.) during the tests,
* Pregnant, parturient or breastfeeding patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2028-06-15 (Estimated)

PRIMARY OUTCOMES:
Analysis of the kinetics of force waves produced at high speed during ballistic movement | 24 Months
  Analysis of the kinetics of force waves produced at high speed during a ballistic movement will make it possible to determine the ability to resume physical activity at a level similar to that before the rupture in the absence of injury (risk = 2.3 / no risk = 0.1).
  Failure to resume physical activity 24 months after ACL surgery is defined by the occurrence of one of the following events:
  * Graft rupture,
  * Contralateral ACL rupture,
  * Decrease of at least 2 points in the Tegner 24 months after cruciate ligament surgery compared to the Tegner before the rupture

SECONDARY OUTCOMES:
Return to physical activity via isokinetic test | 24 Months
  Fitness to resume physical activity via isokinetic test will be determined by quadriceps torque values (>3.0 Nm/kg) and an LSI>90%.
Return to physical activity via the K-STARTS test | 24 Months
  Fitness to resume physical activity via the K-STARTS test will be determined by a total score ≥ 18 points and individual results of the tests comprising the K-START between 2 and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Chantecler, Marseille, France

IPD SHARING:
Plan to Share IPD: No